CLINICAL TRIAL: NCT03644771
Title: Experience With H.P. Acthar Gel Treatment of Patients With Nephrotic Syndrome/Proteinuria Due to Various Etiologies and Its Effect on Podocyte Function
Acronym: Acthar
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Greater Boston Medical Associates (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20150814
Record Dates: First submitted 2018-08-22; First posted 2018-08-23 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Decrease of Proteinuria With H.P. Acthar Gel and Its Effects on Clinical and Podocyte Function
MeSH Terms: interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — one red top tube of blood per month one 50cc urine container per month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Acthar — 4 treatment periods of 3 months each with 20 units biweekly, 40 units biweekly, and 80 units biweekly, with a tapering period to no drug for the fourth 3 month period. Then one year f/u.

SUMMARY:
Patients with proteinuria to start treatment with Acthar and watch a variety of clinical parameters with a goal of decreasing proteinuria between 50-100% over a period of nine months with every 3 months increasing the dose of medication until a decrease of either 50- 100 % of protein excretion is achieved.

In addition addition podocyte function will be assessed monthly by measuring suPar levels, tnf alpha, podocyte/creatinine levels as well as podocyte function studies.

DETAILED DESCRIPTION:
Patients with proteinuria/nephrotic syndrome with albumin/creatinine ratios of 50 or 24 hour urine protein of 500mg or greater will receive increasing doses of H.P. Acthar Gel starting with 20 units weekly or biweekly for 3 months after a one month washout observational period.

The second three month period calls for 40 units biweekly, and the third three month period uses 80 units biweekly observing if the reduction in proteinuria reaches a goal of 50-100%.

Pre study clinical parameters include Cbc diff, cmp, lipid with ldl, cortisol, acth, 24 hour urine for creatinine and protein, urine albumin/creatinine ratio, protein/creatinine ratio, bone density, hgba1c, weight , blood pressure, vital signs, and overall health questionaire. Monthly cbc, cmp, prot/creat, alb/creat ratios, and one red top tube and one 50cc urine container to go to MGH Charlestown for basic podocyte studies. The fourth -3 month observational period will be with tapering to stopping the dose of Acthar and following the same monthly and the pre study parameters.

A second year of observation will continue checking patients every other month for one year to determine the length of protein decrement observed in the first year.

The study will conclude after the second year of drug free followup.

Biomarker studies of podocyte function will be done for the full 2 year period.

Final data analysis will conclude after the 2 year period of observation.

ELIGIBILITY:
Inclusion Criteria:

* patients with proteinuria as above. patients with controlled conditions below are candidates.

Exclusion Criteria:

* uncontrolled hypertension,diabetes mellitus, congestive heart failure, coronary artery disease, peripheral vascular disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18-75 with proteinuria as described.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-01-25 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
level of proteinuria | 2 years
  clinical response and basic science data for podocyte function

CONTACTS AND LOCATIONS:
Locations (1):
- Greater Boston Medical Associates 211 West St., Milford, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Yes if clinically necessary otherwise at end of study